CLINICAL TRIAL: NCT00489385
Title: An Open Label Non-Randomized Trial to Assess Safety and Tolerability of Alb-Interferon Alfa 2b Every Two Weeks With Ribavirin Among HIV/HCV Coinfected Individuals
Brief Title: An Open Label Non-Randomized Dose Escalating Trial to Assess Safety and Tolerability of Alb-Interferon Alfa 2b Every Two Weeks With Ribavirin Among HIV/HCV Coinfected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070001; 07-I-0001
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-01-25

CONDITIONS: HIV Infections; HCV
Keywords: Fibrosis; Viral Kinetics; Hepatotoxicity; Immunity; HIV Infection; Hepatitis C; HCV; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections; Fibrosis; Hepatitis C | interventions — albinterferon alfa-2b; Ribavirin; albuferon

INTERVENTIONS:
Drug: Albinterferon
Drug: Ribavirin
Drug: Albuferon

SUMMARY:
This study will determine if Albumin-linked interferon (Albinterferon alfa-2b) every 2 weeks is safe and tolerated by patients infected by both hepatitis C virus (HCV) and human immunodeficiency virus (HIV). This is a new medication developed for HCV. It may help the immune system fight infections, especially those caused by viruses. Albinterferon alfa-2b appears quite similar to other interferons, in side effects and action in controlling HCV.

Patients ages 18 and older who are infected with HCV genotype 1, are HIV positive, are infected with HCV, and have evidence of HCV-induced liver disease; and who are not pregnant or breast feeding may be eligible for this study. Many visits to NIH over a 76-week period are required. There will be collection of blood and urine, pregnancy test, and tests of HCV in the blood. A liver biopsy is required before start of the study if patients have not had one within 1 year. Another is done at the end of 72 weeks. An eye exam is done before start of the study and repeated later. An optional procedure called automated pheresis is done at the study beginning. Researchers can study patients' immunity to control HCV. Blood is drawn through a needle in an arm vein and spun in a machine to separate the desired blood component. Remaining blood is returned to the patient.

Patients will receive Albinterferon alfa-2b at a dose of 900 mcg every 2 weeks for 48 weeks, by injection under the skin. Ribavirin is given at 1,000 mg or 1,200 mg by mouth twice daily, depending on a patient's weight. Side effects of Albinterferon alfa-2b are fatigue, headache, joint and muscle pain, and sleeplessness. The major side effect of ribavirin is anemia. Visits ranging from week 3 to 44 will determine the safety of Albinterferon alfa-2b and ribavirin and to see effects on reducing the HCV viral load. For weeks 48, 52, 56, 64, 72, and 76, patients will return for a clinic visit and blood tests. At week 72, an abdominal ultrasound and liver biopsy are done. Week 76 includes discussion of biopsy results.

DETAILED DESCRIPTION:
Hepatitis C infection occurs in one-third of all human immunodeficiency virus (HIV)-infected individuals. Liver disease has become more significant among subjects coinfected with HIV and hepatitis C virus (HCV). Several studies have shown that coinfected individuals develop earlier and more severe liver disease. Pegylated interferon alpha with ribavirin (RBV) has become the therapy of choice for HCV among people with HCV alone. However, pegylated interferon with RBV therapy for HIV/HCV coinfected subjects results in only modest cure rates. This is an open-label, non-randomized prospective trial to assess safety and tolerability of Alb-IFN (interferon alpha genetically fused to human serum albumin) 900 mcg every 2 weeks (Q2w) with daily RBV among HIV/HCV coinfected individuals. Twenty-five subjects who are infected with both HIV and HCV and who also have evidence of chronic hepatitis, but who are na ve to anti-HCV treatment, will receive Alb-IFN 900 mcg Q2w together with a standard daily dose of RBV for 48 weeks. These subjects will be monitored for Alb-IFN serum concentration level, HCV viral load, HIV viral load, and CD4 counts, and will undergo a baseline liver biopsy and another optional liver biopsy at the end of 72 weeks. The results of the study will enable us to better delineate the efficacy of Alb-IFN in suppressing the hepatitis C virus in HIV/HCV coinfected subjects. This will be important given the current low cure rate of HCV among HIV coinfected individuals.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 18 years.
  2. Documentation of HIV-1 infection by licensed ELISA test and confirmed by a Western Blot.
  3. Documentation of hepatitis C infection by demonstration of a positive test for hepatitis C antibody and HCV RNA level of 2000 copies/mL or greater.
  4. Histopathologic features consistent with chronic hepatitis C at the time of enrollment. A liver biopsy done for a subject within 24 months prior to his or her participation may be used as the baseline biopsy.
  5. Patients infected with genotype 1.
  6. Patients with CD4+ cell counts greater than 100 cells/mm(3).
  7. Ability to sign the Informed Consent document, and willingness to comply with the study requirements and clinic policies.
  8. Neutrophil count greater than 1000 cells/mm(3).
  9. Platelets greater than 75,000/mm(3).
  10. Hemoglobin greater than 10.5 g/dL.
  11. ALT less than 7 times the NIH upper limit of normal.
  12. Serum lipase less than 1.5 times the NIH upper limit of normal.
  13. Not pregnant or breast-feeding.
  14. If the patient is able to become pregnant, then she must use two effective methods of contraception during the study. Effective contraceptive methods include abstinence, surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap, or sponge, or use of hormonal contraception with an anti-HIV regimen that will not alter metabolism of hormonal contraception. This is advised on the basis of using ribavirin, which may have a potential teratogenic effect on the fetus in pregnant women.
  15. Willingness to not become pregnant until 7 months after completion of ribavirin therapy.
  16. Male subjects who are not documented to be sterile agree to either abstain from intercourse or consistently and correctly use a condom while their female partner (if applicable) agrees to use one of the appropriate medically accepted methods of birth control listed above from the date of screening until 7 months after their last dose of ribavirin.
  17. Patients with a documented addiction are currently in an addiction-free period for at least 6 months and in the clinical judgment of the investigator are not at risk of relapse.
  18. Opioid-dependent patients are in a supervised methadone treatment program.
  19. Need to have a primary doctor outside of OP8 or as part of the OP8 training clinic who will be taking care of the patients for their HIV infection and liver disease.
  20. Willing to designate a person for durable power of attorney on the NIH form for medical research and medical care purposes at the NIH Clinical Center.
  21. Able to learn to safely inject medication Alb-IFN subcutaneously or be able to find another person or a clinic to inject the medication for him/her.
  22. Willingness to abstain from alcohol use during the trial.
  23. Willingness to allow stored blood or tissue samples to be used in the future for studying HIV disease and immune function.
  24. Willingness to permit HLA typing to be performed.

EXCLUSION CRITERIA:

1. Patient cannot be on other experimental therapies (including expanded access/compassionate use of antiretrovirals) during his/her participation in this protocol.
2. Patients cannot have used interferon or peginterferon previously for the treatment of hepatitis C.
3. Mixed genotypes (e.g., 1/2, 1/4). Mixed genotype 1a/1b will be enrolled.
4. Liver histology which, in the opinion of Clinical Center pathologist, is consistent with any other co-existent cause of chronic liver disease as defined as: chronic hepatitis B with positive HBsAg autoimmune hepatitis with a positive ANA greater than 1 unit or positive anti mitochondrial antibody greater than 1 unit; cholestatic disease with persistent elevation of alkaline phosphatase; primary biliary cirrhosis or sclerosing cholangitis; Wilson's disease; alpha-1-antitrypsin deficiency; steatohepatitis (alcoholic or non alcoholic) with marked steatosis, many Mallory bodies, or extensive zone 3 periportal fibrosis.
5. Hemochromatosis or secondary iron overload as defined by (1) an elevated serum ferritin or an iron saturation (serum iron/IBC times 100%) of greater than 50%, and (2) presence of 3+ or more stainable iron on liver biopsy according to the study pathologist. Those subjects with, or a history of previous phlebotomy for iron overload will undergo HFE genetic counseling and those with a positive HFE genetic test demonstrating homozygosity for C282Y and H63D are not eligible. Those who have compound heterozygosity to C282Y and H63D are also not eligible.
6. For patients with cirrhosis, a Child Turcotte Pugh score greater than 7.
7. PT-INR greater than 2 or history of hemophilia or known history of Vitamin K deficiency or use of anticoagulants.
8. Organ transplant recipient other than cornea or hair transplant.
9. Estimated Creatinine clearance (eGFR) less than 50 mL/min.
10. A serum alpha-fetoprotein level (greater than 20 ng/mL, unless the subject has a negative ultrasound before enrollment.
11. For patients with history of diabetes mellitus, a HbA1C less than or equal to 7.5% and for those with a fasting blood glucose level of greater than 140mg/dL, a HbA1C of less than or equal to 7.5%.
12. Coexisting neoplastic disease except for Kaposi's sarcoma, any non-metastatic skin cancer that has been resected, or non-metastatic cervical or anal cancer that has been resected.
13. Severe cardiac disease (Grade 3 or more congestive cardiac failure, symptomatic coronary artery disease, significant arrhythmias, uncontrolled hypertension).
14. Severe chronic pulmonary disease with functional impairment or a DLCO less than or equal to 50% at baseline.
15. Severe psychiatric disorder that would interfere with the adherence to protocol requirements.
16. Preexisting autoimmune disorders including inflammatory bowel diseases, psoriasis, and optic neuritis.
17. Preexisting uncontrolled seizure disorder defined as one episode of seizure within the past 2 years.
18. Chronic pancreatitis.
19. Severe retinopathy as determined by the ophthalmologist.
20. Hemoglobinopathy (e.g., Thalassemia, sickle cell disease).
21. Currently taking didanosine or d4T as part of antiretroviral regimen.
22. Direct bilirubin greater than or equal to 0.6 mg/dL.
23. Concurrent use of any immunosuppressive therapy, including systemic steroids (prednisone equivalent of greater than 10 mg/day) for a duration of six weeks or more within six months prior to enrollment.
24. Concurrent use of fluticasone and high dose ritonavir (600mg t.i.d).
25. Chronic viral hepatitis of any other etiology other than hepatitis C.
26. Active systemic infections other than hepatitis C and HIV.
27. Liver disease caused by reasons other than hepatitis C, like HBV, HDV, Wilson's disease, hemochromatosis, autoimmune hepatitis (ANA greater than 1 unit) except history of drug-associated hepatitis with discontinuation of the causative agent.
28. Hepatic mass suggestive of hepatocellular carcinoma as detected by ultrasound scan.
29. Alcohol or substance abuse within the past 6 months that potentially could interfere with patient compliance.
30. Concomitant use of amphetamines, barbiturates, cocaine, ganciclovir, isoniazid, opiates, pyrazinamide, rifabutin, rifampin/rifampicin, thalidomide, and theophylline.
31. History of esophageal varices.
32. Any systemic illness that will make it unlikely that the subject will be able to return to NIH for the required study visits.
33. Evidence of gastrointestinal malabsorption, chronic nausea, or vomiting.
34. Male partners of pregnant women.
35. Pregnant women.
36. Breastfeeding women.
37. Hypersensitivity to interferon products or ribavirin.
38. Received silymarin (milk thistle) or glycyrrhizin within 28 days prior to Day 0.
39. Received Sho-saiko-to (SST) within 28 days prior to Day 0.
40. Received any other experimental agent within 28 days prior to Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-06-18; Primary Completion 2011-03-15 (Actual); Study Completion 2011-03-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of two doses of Albinterferon alpha 2b with ribavirin.

SECONDARY OUTCOMES:
Histologic, virologic responses to Albinterferon alpha 2b and ribavirin

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alter MJ, Mast EE. The epidemiology of viral hepatitis in the United States. Gastroenterol Clin North Am. 1994 Sep;23(3):437-55. PMID 7989088
- [Background] Seeff LB, Buskell-Bales Z, Wright EC, Durako SJ, Alter HJ, Iber FL, Hollinger FB, Gitnick G, Knodell RG, Perrillo RP, et al. Long-term mortality after transfusion-associated non-A, non-B hepatitis. The National Heart, Lung, and Blood Institute Study Group. N Engl J Med. 1992 Dec 31;327(27):1906-11. doi: 10.1056/NEJM199212313272703. PMID 1454085
- [Background] Koretz RL, Abbey H, Coleman E, Gitnick G. Non-A, non-B post-transfusion hepatitis. Looking back in the second decade. Ann Intern Med. 1993 Jul 15;119(2):110-5. doi: 10.7326/0003-4819-119-2-199307150-00003. PMID 8512159